CLINICAL TRIAL: NCT06063382
Title: Extended Time on Exams as an Accommodation at First Level of Higher Education: A Randomized Controlled Study
Brief Title: Extra Time on Brazilian College Level Exam for Students With and Without ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0458; 64785722.0.0000.5327 (Other: Ethics Committee - Brazilian Government (CEP/Conep))
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Extended time; Academic test Performance; Academic Achievement; Neuropsychological Testing; Cognitive Function
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants will be assigned either to the "ADHD group" or "non-ADHD group" based on diagnosis. Both groups will receive the same intervention, which is to perform three academic exams based on the Brazilian National High School Exam (ENEM) under three different time conditions (40 minutes, 50 minutes and 60 minutes). The order in which they will perform each exam and with which time condition will be randomized.
  In order to emulate real-life conditions in which students compete for college entry and motivate them, the participants will be competing for valuable prizes (ebook readers).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD group (Experimental): Participants with Attention Deficit Disorder/Hyperactivity (ADHD) diagnosis who will take three equivalent academic exams, having 40 minutes (standard time), 50 minutes (25% increase) and 60 minutes (50% increase) to complete the exam.
  Interventions: Behavioral: Extended time 25%; Behavioral: Extended time 50%
- Control group (Active Comparator): Participants without Attention Deficit Disorder/Hyperactivity (ADHD) diagnosis who will take three equivalent academic exams, having 40 minutes (standard time), 50 minutes (25% increase) and 60 minutes (50% increase) to complete the exam.
  Interventions: Behavioral: Extended time 25%; Behavioral: Extended time 50%

INTERVENTIONS:
Behavioral: Extended time 25% — Considering a standard time of 40 minutes, participants will receive 50 minutes to complete the exam.
Behavioral: Extended time 50% — Considering a standard time of 40 minutes, participants will receive 50 minutes to complete the exam.

SUMMARY:
Standardized tests such as the Scholastic Aptitude Test (SAT) and the brazilian National High School Exam (ENEM) give more time for students with Attention Deficit and Hyperactivity Disorders (ADHD) to complete the exam. The goal of this study is to find out if giving students with ADHD more time on tests actually helps them. Additionally, the research aims to find out if more time helps students without ADHD too or not, or even if it only helps students with certain traits.

DETAILED DESCRIPTION:
Initially, the participants of this study will fill out forms and questionnaires online. Then, they will go through a psychiatric evaluation, where they will talk to a psychiatrist, and neuropsychological testing, where they will do some mental activities. Later on, they will do a mock test of the ENEM, with and without extra time.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian citizen;
* Planing to participate in college-entry standardized tests (ENEM, Vestibulares);

Exclusion Criteria:

* Medical condition and/or disability that may hinder the neuropsychological testing;
* Intelligence Quotient (IQ) lower than 80;
* Psychotic disorders, bipolar disorders, current moderate or severe depressive episode, suicide risk, autism spectrum disorders, learning disabilities.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Test Scores Under Three Time-Limited Testing Conditions. | During a two-hour-and-a-half intervention.
  Test performance measured by the proportion of correct answers weighted according to the Item Response Theory.

SECONDARY OUTCOMES:
Between-Group Difference in Change from Baseline in Test Scores Under Three Time-Limited Testing Conditions (ADHD vs. Non-ADHD Participants). | During a two-and-a-half-hour intervention.
  Test performance measured by the proportion of correct answers weighted according to the Item Response Theory.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto Paim Rohde, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Online questionnaires — https://redcap.link/ognsz470